CLINICAL TRIAL: NCT00967577
Title: 177Lu Radiolabeled Monoclonal Antibody HuJ591-GS (177Lu-J591) in Patients With Nonprostate Metastatic Solid Tumors: A Pilot Study
Brief Title: 177Lu-J591 Antibody in Patients With Nonprostate Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0902010212
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Kidney Cancer; Head and Neck Cancer; Breast Cancer; Non-small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Ovarian Cancer; Esophageal Cancer; Gliomas
MeSH Terms: conditions — Kidney Neoplasms; Head and Neck Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms; Glioma | interventions — J591 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- J591 (Experimental)
  Interventions: Drug: 177Lu-J591

INTERVENTIONS:
Drug: 177Lu-J591 — 70 mCi/m2 of 177Lu-J591 will be administered on Day 1.
  Other Names: monoclonal antibody J591

SUMMARY:
The purpose of this study is to evaluate changes in tumor blood flow and disease response to the investigation agent, 177Lu-J591.

DETAILED DESCRIPTION:
177Lu-J591 is made up of two compounds called J591 and 177Lutetium (177Lu) that are joined together by a connecting molecule called "DOTA". J591 is a monoclonal antibody, or a type of protein. 177Lu is a radioactive molecule that is being tested for the possible treatment of cancer when joined to monoclonal antibodies. J591 attaches to a protein called prostate specific membrane antigen (PSMA) found in the body. PSMA is mostly found in normal and cancerous prostate cells. In addition, however, PSMA has also been found on the vasculature (blood vessels) that supply multiple types of cancer including colorectal, kidney, bladder, head and neck, breast, non-small cell lung, pancreas, ovary, esophagus and gliomas.

We hope that 177Lu-J591 will seek out blood vessels that supply these tumors and deliver a dose of radiation (from the 177Lu molecule) to the areas of cancer, without affecting target blood vessel that are not associated with the cancer.

Zirconium-89 (89Zr) is a radioactive tracer that allows special scans to be performed prior to administration of the study drug to determine where the antibody goes in the body and to screen the tumor's blood vessels to see if they attract J591. Again, DOTA is used to join the radioactive material to J591. 89Zr-J591 is not being given to treat cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically, or cytologically documented, advanced stage, malignant adult solid tumors (except prostate cancer) that are refractory to, or recurrent from, standard therapy or for which no curative standard therapy exists. This will include, but is not limited to patients with cancers of the kidney, urothelium, head and neck, breast, non-small cell lung, colorectal, pancreas, ovary, esophagus and gliomas.
* Metastatic or recurrent solid tumor malignancy defined by abnormal CT, MRI, PET scan, CXR and/or bone scan
* Progressive disease manifest by: Development of new lesions or an increase in size of preexisting lesions on imaging study or by physical examination.
* Subjects must have recovered from the acute toxicities of any prior therapy, and not received chemotherapy, radiation therapy or other investigational anticancer therapeutic drug for at least 4 weeks prior to J591 administration in this trial
* All subjects must have archived or current tissue (from a primary or metastatic focus) available for PSMA determination.
* Subjects on bisphosphonate therapy or denosumab must be on a stable dose and must have started therapy > 4 weeks prior to protocol therapy.
* Subjects will be informed as to the potential risk of procreation while participating on this trial and will be advised to use effective contraception during the entire study period. Females of child-bearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Use of platelet transfusions within 4 weeks of treatment.
* Use of hematopoietic growth factors within 4 weeks of treatment.
* Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of treatment.
* Prior radiation therapy encompassing >25% of skeleton.
* Prior treatment with 89Strontium or 153Samarium containing compounds (e.g. Metastron®, Quadramet®)
* Platelet count <150,000/mm3 or history of platelet count abnormality or dysfunction.
* Absolute neutrophil count (ANC) <2,000/mm3
* Hematocrit <30 percent or Hemoglobin < 10 g/dL
* Abnormal coagulation profile (PT or INR, PTT) > 1.3x upper limit of normal (ULN) unless on therapeutic anticoagulation
* Serum creatinine > 2x ULN
* AST (SGOT) >2.5x ULN
* Bilirubin (total) >1.5x ULN; subjects with known Gilbert's syndrome are eligible if direct bilirubin is within institutional normal limits
* Active serious infection
* Active angina pectoris or NY Heart Association Class III-IV
* ECOG Performance Status > 2
* Deep vein thrombosis and/or pulmonary embolus within 1 month of enrollment.
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.
* Prior investigational therapy (medications or devices) within 4 weeks of treatment.
* Known history of HIV.
* Known leukemia or myelodysplastic syndrome
* Prior allergic reaction to Gadolinium contrast.
* Life expectancy < 3 months
* If alternative treatments are available, metastatic disease should not be progressing so as to anticipate the necessity of urgent treatment within 12 weeks of enrollment based on clinical assessment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in tumor perfusion as based on Dynamic Contrast Enhanced (DCE)-MRI study | Performed after administration of 177LuJ591 between Day 6-9 and on Day 29.
Change in tumor perfusion based on changes in cellularity as assessed using Diffusion-weighted imaging (DWI) | Performed after administration of 177LuJ591 between Day 6-9 and on Day 29.

SECONDARY OUTCOMES:
Changes in response rate using Response evaluation criteria in solid tumors (RECIST) Criteria | Objective response will be evaluated from changes in baseline to Day 99 and repeated every 3 months until radiographic progression of disease.
  Through RECIST criteria, objective response will be evaluated by taking into account the measurement of the longest diameter only for all target lesions on CT scans as well as normalization of serum tumor markers (if applicable).
Change in the number of subjects who achieve Progression Free Survival | Day 58 after administration with 177Lu-J591 and repeated every 3 months until radiographic progression of disease
  Progression free survival is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. This will be calculated from the time of treatment (day of 177Lu-J591 infusion) until radiographic progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No